CLINICAL TRIAL: NCT00042939
Title: Phase II Trial of Irinotecan/Docetaxel for Advanced Pancreatic Cancer, With Randomization Between Irinotecan/Docetaxel and Irinotecan/Docetaxel Plus C225 a Monoclonal Antibody to the Epidermal Growth Factor Receptor (EGF-r)
Brief Title: Irinotecan and Docetaxel With or Without Cetuximab in Treating Patients With Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000069486; U10CA021115 (NIH); E8200 [ECOG] (Other: Eastern Cooperative Oncology Group (ECOG))
Record Dates: First submitted 2002-08-05; First posted 2003-01-27 (Estimated); Results first posted 2011-07-19 (Estimated); Last update posted 2023-07-06 (Actual); Status verified 2023-06

CONDITIONS: Pancreatic Cancer
Keywords: pancreatic cancer; metastatic pancreatic cancer; EGF-r; irinotecan; docetaxel; cetuximab
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Cetuximab; Docetaxel; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Irinotecan/Docetaxel (Active Comparator): Docetaxel was administered intravenously over 60 minutes at a dose of 35 mg/m². Docetaxel was diluted in 100-150 ml of infusion solution. After the completion of the docetaxel infusion, irinotecan was administered intravenously over 30 minutes at a dose of 50 mg/m².
  Chemotherapy was administered once a week (days 1, 8, 15, 22) for 4 consecutive weeks followed by 2 weeks rest. This constituted a cycle of treatment. Patients were evaluated after 2 cycles.
  Interventions: Drug: docetaxel; Drug: irinotecan hydrochloride
- Irinotecan/Docetaxel/Cetuximab (Experimental): Patients received Cetuximab intravenously once a week for 6 weeks. On day 1 of cycle 1 only, an initial dose of 400 mg/m² (over 120 minutes) was administered. Thereafter, a once-a-week maintenance dose of 250 mg/m² (infused over 60 minutes), was given. The infusion rate never exceeded 5 ml/minute.
  On the day of the initial dose, the administration of Cetuximab was followed by the administration of docetaxel, after a 60-minute observation period. (The observation period was 30 minutes following maintenance doses.) Docetaxel was administered intravenously over 60 minutes at a dose of 35 mg/m². Docetaxel was diluted in 100-150 ml of infusion solution. After the completion of the docetaxel infusion, irinotecan was administered intravenously over 30 minutes at a dose of 50 mg/m².
  Chemotherapy was administered once a week (days 1, 8, 15, 22) for 4 consecutive weeks followed by 2 weeks rest. Cetuximab was administered once a week for 6 consecutive weeks. A cycle of treatment was 6 weeks.
  Interventions: Biological: cetuximab; Drug: docetaxel; Drug: irinotecan hydrochloride

INTERVENTIONS:
Biological: cetuximab — Patients received cetuximab intravenous infusions, via infusion pump or syringe pump, once a week for 6 weeks.
  Other Names: Erbitux; C225
  Arms: Irinotecan/Docetaxel/Cetuximab
Drug: docetaxel — Docetaxel was administered intravenously over 60 minutes at a dose of 35 mg/m² once a week (days 1, 8, 15, 22) for 4 consecutive weeks followed by 2 weeks rest. Docetaxel was diluted in 100-150 ml of infusion solution.
  Other Names: Taxotere
Drug: irinotecan hydrochloride — After the completion of the docetaxel infusion, irinotecan was administered intravenously over 30 minutes at a dose of 50 mg/m² once a week (days 1, 8, 15, 22) for 4 consecutive weeks followed by 2 weeks rest.
  Other Names: Camptosar

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Monoclonal antibodies such as cetuximab can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Combining chemotherapy with cetuximab may kill more tumor cells.

PURPOSE: This randomized phase II trial is studying giving irinotecan and docetaxel together with cetuximab to see how well it works compared to irinotecan and docetaxel alone in treating patients with metastatic pancreatic cancer .

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of irinotecan and docetaxel with or without cetuximab, in terms of objective response rate, in patients with metastatic adenocarcinoma of the pancreas.
* Determine the time to progression and overall survival of patients treated with these regimens.
* Determine the proportion of patients with tumors that overexpress epidermal growth factor receptor.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm A: Patients receive docetaxel IV over 1 hour and irinotecan IV over 30 minutes weekly on days 1, 8, 15, and 22.
* Arm B: Patients receive docetaxel and irinotecan as in arm A. Patients also receive cetuximab IV over 1-2 hours on days 1, 8, 15, 22, 29, and 36.

Courses repeat in both arms every 6 weeks in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 2 years, every 6 months for 1 year, and then periodically thereafter.

PROJECTED ACCRUAL: A total of 92 patients (46 per treatment arm)

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic adenocarcinoma of the pancreas
* Sufficient tumor tissue from fine needle aspiration, core biopsy, or open biopsy available for epidermal growth factor receptor testing
* At least 1 unidimensionally measurable primary or metastatic lesionge
* Age of 18 and over
* ECOG performance status 0-1
* Negative pregnancy test
* Fertile patients must use effective contraception
* Creatinine clearance > 60 mL/min
* LVEF normal
* Absolute neutrophil count > 1,500/mm^3
* Platelet count > 100,000/mm^3
* Bilirubin ≤ upper limit of normal (ULN)*
* SGOT or SGPT and alkaline phosphatase must meet the criteria for 1 of the following*:

  * SGOT or SGPT ≤ 2.5 times ULN AND alkaline phosphatase ≤ ULN
  * SGOT or SGPT ≤ 1.5 times ULN AND alkaline phosphatase > ULN but ≤ 2.5 times ULN
  * SGOT or SGPT ≤ ULN AND alkaline phosphatase > 2.5 but ≤ 4 times ULN

NOTE: *Percutaneous stenting or endoscopic retrograde cholangiopancreatography may be used to normalize liver function tests

Exclusion Criteria:

* History of uncontrolled arrhythmias
* History of congestive heart failure
* History of uncontrolled angina pectoris
* Prior chemotherapy
* Pre-existing neuropathy ≥ grade 2
* Prior hypersensitivity to polysorbate 80
* Pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2003-12-09 (Actual); Primary Completion 2009-06 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara A. Burtness, MD, Study Chair — Fox Chase Cancer Center

REFERENCES:
- [Result] Burtness BA, Powell ME, Berlin JD, et al.: Phase II ECOG trial of irinotecan/docetaxel with or without cetuximab in metastatic pancreatic cancer: updated survival and CA19-9 results. [Abstract] J Clin Oncol 26 (Suppl 15): A-4642, 2008.
- [Result] Burtness BA, Powell M, Berlin J, et al.: Phase II trial of irinotecan/docetaxel for advanced pancreatic cancer with randomization between irinotecan/docetaxel and irinotecan/docetaxel plus C225, a monoclonal antibody to the epidermal growth factor receptor (EGF-r) : Eastern Cooperative Oncology. [Abstract] J Clin Oncol 25 (Suppl 18): A-4519, 2007.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: E8200 opened to accrual on 7/31/2003, accrued its first patient on 12/9/2003, and was suspended on 12/2/2004 for evaluation of response and toxicity. Arm B was reactivated on 7/12/2005 after meeting the response criteria; Arm A was reactivated on 11/23/2005. Arm B and Arm A closed to accrual on 4/17/2006 and 8/23/2006, respectively, after meeting the accrual goal.
Groups:
- Arm A: Irinotecan/Docetaxel: Docetaxel was administered intravenously over 60 minutes at a dose of 35 mg/m². Docetaxel was diluted in 100-150 ml of infusion solution. After the completion of the docetaxel infusion, irinotecan was administered intravenously over 30 minutes at a dose of 50 mg/m².
  Chemotherapy was administered once a week (days 1, 8, 15, 22) for 4 consecutive weeks followed by 2 weeks rest. This constituted a cycle of treatment. Patients were evaluated after 2 cycles.
- Arm B: Irinotecan/Docetaxel/Cetuximab: Patients received Cetuximab intravenously once a week for 6 weeks. On day 1 of cycle 1 only, an initial dose of 400 mg/m² (over 120 minutes) was administered. Thereafter, a once-a-week maintenance dose of 250 mg/m² (infused over 60 minutes), was given. The infusion rate never exceeded 5 ml/minute.
  On the day of the initial dose, the administration of Cetuximab was followed by the administration of docetaxel, after a 60-minute observation period. (The observation period was 30 minutes following maintenance doses.) Docetaxel was administered intravenously over 60 minutes at a dose of 35 mg/m². Docetaxel was diluted in 100-150 ml of infusion solution. After the completion of the docetaxel infusion, irinotecan was administered intravenously over 30 minutes at a dose of 50 mg/m².
  Chemotherapy was administered once a week (days 1, 8, 15, 22) for 4 consecutive weeks followed by 2 weeks rest. Cetuximab was administered once a week for 6 consecutive weeks. A cycle of treatment was 6 weeks.
Period: Overall Study
Arm/Group | Arm A: Irinotecan/Docetaxel | Arm B: Irinotecan/Docetaxel/Cetuximab
Started | 48 | 46
Treated | 46 | 45
Eligible and Began Protocol Therapy | 44 | 43
Patients With EGFR Results Available | 30 | 31
Completed | 24 | 25
Not Completed | 24 | 21
Not completed — Adverse Event | 6 | 7
Not completed — Death | 3 | 2
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Other disease | 1 | 0
Not completed — Ineligible | 2 | 2
Not completed — Deterioration of health | 3 | 4
Not completed — QOL diminished | 1 | 0
Not completed — Rising ca 19-9 | 1 | 0
Not completed — Patient non-compliance | 1 | 0
Not completed — Still on treatment | 1 | 0
Not completed — Treatment break > 4 weeks | 0 | 1
Not completed — Did not start treatment | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Irinotecan/Docetaxel | Arm B: Irinotecan/Docetaxel/Cetuximab | Total
Number analyzed (Participants) | 44 | 43 | 87
Age, Continuous [Median (Full Range); unit: years] — Age of eligible patients who began treatment.
  years | 60.2 [41.0 to 77.1] | 60.6 [41.0 to 74.2] | 60.4 [41.0 to 77.1]
Sex: Female, Male [Count of Participants; unit: Participants] — Gender of eligible patients who began treatment.
  Participants
    Female | 20 | 6 | 26
    Male | 24 | 37 | 61

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Objective Response Evaluated by RECIST (Solid Tumor Response Criteria)
Description: Per RECIST criteria, Complete response (CR)= disappearance of all target and nontarget lesions Partial response (PR)= >=30% decrease in the sum of the longest diameters of target lesions from baseline, and persistence of one or more non-target lesion(s) and/or the maintenance of tumor marker level above the normal limits.
  Objective response = CR + PR
Time Frame: Assessed every 12 weeks until progression
Population: Eligible patients who began treatment were included in the analysis.
Measure: Number (90% Confidence Interval); unit: Proportion of participants
Arm/Group | Arm A: Irinotecan/Docetaxel | Arm B: Irinotecan/Docetaxel/Cetuximab
Number analyzed (Participants) | 44 | 43
Proportion of participants | 0.045 [0.015 to 0.184] | 0.07 [0.024 to 0.198]

2. Secondary Outcome: Progression-free Survival
Description: Progression-free survival was defined as the shorter of:
  1. The time from registration to progression. or
  2. The time from registration to death without documentation of progression given that the death occured within 4 months of the last disease assessment without progression (or registration, whichever is more recent).
  Progression is defined as at least a 20% increase in the sum of the longest diameters of target lesions, taking as reference the smallest sum longest diameter recorded since the baseline measurements, or the appearance of one or more new lesion(s) or unequivocal progression of existing nontarget lesions.
Time Frame: Assessed every 3 months for 2 years and then every 6 months for 1 year
Population: Eligible patients who began treatment.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Arm A: Irinotecan/Docetaxel | Arm B: Irinotecan/Docetaxel/Cetuximab
Number analyzed (Participants) | 44 | 43
months | 3.9 [2.4 to 5.0] | 4.5 [2.7 to 5.6]

3. Secondary Outcome: Overall Survival
Description: Overall survival was defined as time from registration to death from any cause.
Time Frame: Assessed every 3 months for 2 years and then every 6 months for 1 year
Population: Eligible patients who began treatment.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Arm A: Irinotecan/Docetaxel | Arm B: Irinotecan/Docetaxel/Cetuximab
Number analyzed (Participants) | 44 | 43
months | 6.5 [5.6 to 9.9] | 5.3 [4.5 to 9.4]

4. Secondary Outcome: Epidermal Growth Factor Receptor (EGFR) Status
Description: EGFR expression was be evaluated by staining 5-micron paraffin sections of tumor biopsies with anti-EGFR clone 2-18C9 (DAKO Corporation, Carpinteria, CA) using an indirect immunoperoxidase technique according to the instructions provided by DAKO. In brief, this includes an antigen retrieval pretreatment, the blocking of endogenous peroxidase activity, incubation with anti-EGFR antibody or a negative reagent control, staining with a detection system, visualization, and coverslipping.
Time Frame: Original tumor tissue samples submitted within one month of patient randomization
Population: Eligible and treated patients with EGFR stain results available.
Measure: Number; unit: participants
Arm/Group | Arm A: Irinotecan/Docetaxel | Arm B: Irinotecan/Docetaxel/Cetuximab
Number analyzed (Participants) | 30 | 31
participants
  Positive | 29 | 30
  Negative | 1 | 1

5. Secondary Outcome: Proportion of Patients With Thromboembolic Events
Description: To determine the rate of thromboembolic events in this population when prophylactic enoxaparin sodium is administered.
Time Frame: Assessed every 6 weeks while on treatment and for 30 days after the end of treatment
Population: Eligible and treated patients
Measure: Number (90% Confidence Interval); unit: Proportion of participants
Arm/Group | Arm A: Irinotecan/Docetaxel | Arm B: Irinotecan/Docetaxel/Cetuximab
Number analyzed (Participants) | 44 | 43
Proportion of participants | 0 [0.0 to 0.066] | 0.023 [0.001 to 0.106]

ADVERSE EVENTS:
Time Frame: Assessed every 6 weeks while on treatment and for 30 days after the end of treatment.
Arm/Group | Arm A: Irinotecan/Docetaxel | Arm B: Irinotecan/Docetaxel/Cetuximab
Serious Adverse Events (participants affected / at risk) | 35/46 | 36/45
Other Adverse Events (participants affected / at risk) | 46/46 | 45/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Irinotecan/Docetaxel (N=46) | Arm B: Irinotecan/Docetaxel/Cetuximab (N=45)
Allergic Reaction (Immune system disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 4 | 9
Leukopenia (Investigations) | 12 | 13
Lymphopenia (Investigations) | 0 | 1
Neutropenia (Investigations) | 10 | 13
Transfusion: pRBCs (Blood and lymphatic system disorders) | 5 | 2
Supraventricular Arrhythmias (Cardiac disorders) | 0 | 1
Edema (General disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 3
Pericardial Effusion/Pericarditis (Cardiac disorders) | 0 | 1
Thrombosis/Embolism (Vascular disorders) | 0 | 1
Fatigue (General disorders) | 10 | 8
Fever (General disorders) | 1 | 1
Weight Loss (Investigations) | 0 | 1
DIC (Disseminated Intravascular Coagulation) (Blood and lymphatic system disorders) | 1 | 0
Rash/Desquamation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin-Other (Skin and subcutaneous tissue disorders) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 8 | 4
Ascites (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Ddhydration (Metabolism and nutrition disorders) | 4 | 8
Dysphagia (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 14 | 9
Stomatitis (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 6 | 9
Diarrhea w/o Prior Colostomy (Gastrointestinal disorders) | 14 | 21
GI -Other (Gastrointestinal disorders) | 0 | 1
Hematuria (Renal and urinary disorders) | 0 | 1
Melena/GI Bleeding (Gastrointestinal disorders) | 0 | 2
Alkaline Phosphatase Increased (Investigations) | 3 | 3
Bilirubin Increased (Investigations) | 1 | 1
AST Increased (Investigations) | 3 | 1
ALT Increased (Investigations) | 3 | 3
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 | 2
Infection w/ Grade 3 or 4 Neutropenia (Infections and infestations) | 2 | 3
Infection w/ Unknown ANC (Infections and infestations) | 1 | 1
Infection w/o Neutropenia (Infections and infestations) | 3 | 3
Infection -Other (Infections and infestations) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 3 | 5
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 3
Hyponatremia (Metabolism and nutrition disorders) | 2 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 1
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 3 | 0
Dizziness/Lightheadedness (Nervous system disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0
Anxiety/Agitation (Psychiatric disorders) | 1 | 0
Neuropathy-Motor (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Conjunctivitis (Eye disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 2 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain-Other (General disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Syndromes-Other (General disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Irinotecan/Docetaxel (N=46) | Arm B: Irinotecan/Docetaxel/Cetuximab (N=45)
Anemia (Blood and lymphatic system disorders) | 40 | 41
Leukopenia (Investigations) | 33 | 31
Neutropenia (Investigations) | 24 | 24
Thrombocytopenia (Investigations) | 11 | 6
Edema (General disorders) | 5 | 5
Hypotension (Vascular disorders) | 2 | 3
Fatigue (General disorders) | 32 | 31
Fever (General disorders) | 6 | 6
Rigors/ Chills (General disorders) | 7 | 3
Weight Loss (Investigations) | 15 | 16
Alopecia (Skin and subcutaneous tissue disorders) | 25 | 22
Dry Skin (Skin and subcutaneous tissue disorders) | 4 | 8
Nail Changes (Skin and subcutaneous tissue disorders) | 8 | 7
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 4
Rash/Desquamation (Skin and subcutaneous tissue disorders) | 4 | 30
Skin-Other (Skin and subcutaneous tissue disorders) | 3 | 10
Hot Flashes (Vascular disorders) | 2 | 3
Anorexia (Metabolism and nutrition disorders) | 22 | 25
Constipation (Gastrointestinal disorders) | 7 | 9
Dehydration (Metabolism and nutrition disorders) | 7 | 3
Dyspepsia (Gastrointestinal disorders) | 5 | 4
Mouth Dryness (Gastrointestinal disorders) | 4 | 8
Nausea (Gastrointestinal disorders) | 23 | 28
Stomatitis (Gastrointestinal disorders) | 8 | 21
Taste Disturbance (Nervous system disorders) | 6 | 15
Vomiting (Gastrointestinal disorders) | 25 | 20
Diarrhea w/o Prior Colostomy (Gastrointestinal disorders) | 27 | 29
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 7
Alkaline Phosphatase Increased (Investigations) | 19 | 21
Bilirubin Increased (Investigations) | 6 | 14
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 | 4
AST Increased (Investigations) | 6 | 16
ALT Increased (Investigations) | 10 | 23
Infection w/o Neutropenia (Infections and infestations) | 5 | 5
Hyperglycemia (Metabolism and nutrition disorders) | 7 | 5
Hypocalcemia (Metabolism and nutrition disorders) | 3 | 5
Hypokalemia (Metabolism and nutrition disorders) | 1 | 4
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 9
Hyponatremia (Metabolism and nutrition disorders) | 3 | 6
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 6 | 1
Dizziness/Lightheadedness (Nervous system disorders) | 2 | 6
Insomnia (Psychiatric disorders) | 1 | 3
Depression (Psychiatric disorders) | 1 | 3
Neuropathy-Motor (Nervous system disorders) | 3 | 2
Neuropathy-Sensory (Nervous system disorders) | 7 | 12
Tearing (Eye disorders) | 5 | 2
Abdominal Pain (Gastrointestinal disorders) | 11 | 7
Headache (Nervous system disorders) | 3 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 9
Hiccoughs (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Creatinine Increased (Investigations) | 4 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No